CLINICAL TRIAL: NCT01874457
Title: A Serological Study of Measles, Mumps and Rubella in Children 12 to 23 Months Vaccinated With MMR (Measles, Mumps and Rubella) in Health Centers Where a Phase III Study Should be Conducted
Brief Title: Serological Study in Children 12 to 23 Months Vaccinated With MMR (Measles, Mumps and Rubella)
Status: Completed | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN/002/2008
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Mumps; Rubella; Measles
MeSH Terms: conditions — Mumps; Rubella; Measles | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MMR (Mumps, Measles and Rubella) — MMR (Mumps, Measles and Rubella)

SUMMARY:
On a previous study conducted in Brazil. The MMR vaccine from 2 different producers had a mumps seroconversion much lower (71%) than the expected 95%, according to the package insert. This could indicate that a substantial proportion of children was not protected after MMR dose.

DETAILED DESCRIPTION:
Given the above and considering: (1) future clinical study with the MMR vaccine produced entirely in Bio-Manguinhos/Fiocruz from technology transfer from GlaxoSmithKline (GSK), (2) the importance to the National Immunization Program (NIP) to provide the population a MMR vaccine to ensure high protection against mumps, similar to what occurs with measles and rubella components, it was considered essential to conduct a preliminary immunogenicity assessment of the MMR vaccine produced by BioManguinhos.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes;
* Age between 12 months to 23 months and 29 days;
* Child in good health, with no significant past medical history;
* Have completed blood sampling before vaccination;
* Have not been vaccinated with MMR.
* Agreement by parents/tutors with the child's participation in the study and signing of the Informed Consent Form (ICF);
* Parents/Tutors provide name, address, telephone number and other information for the contact if necessary;
* Parents/Tutors able to understand the risks of the experiment, although minimal;
* Parents/Tutors able to understand and sign the informed consent form.
* Availability of return for collecting post-vaccination samples.

Exclusion criteria:

* Children with a history of measles, rubella and / or mumps.
* Having received MMR vaccine previously, as documented in vaccination card.
* Having received a transfusion of blood or blood products, including immunoglobulins, within last 12 months.
* Skin lesions at sites of venipuncture.
* Child subject to abnormal bleeding after injections.
* Use within 6 months of corticosteroids (excluding topical or aerosol) and immunosuppressants.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 12-23 months and 29 days old, in the routine of PNI in health units in the city of Rio de Janeiro.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Immunoresponse after first dose | 42 days
  Assess the immunoresponse for measles, mumps and rubella after vaccination with MMR in children 12-23 months and 29 days old, in the routine of National Immunization Program (NIP) in health units in the city of Rio de Janeiro.

SECONDARY OUTCOMES:
Immunoresponse after revaccination | 42 days
  To evaluate the immunoresponse after revaccination of children who did not seroconvert for any of the three components of the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Glória Regina da Silva e Sá, Doctorate, Principal Investigator — Immunobiological Technology Institute (Bio-Manguinhos)
Locations (1):
- Bio-Manguinhos/Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil